CLINICAL TRIAL: NCT03270657
Title: Scalar Closed-Loop STN/GPi DBS Based on Evoked and Spontaneous Potentials (Intraoperative Studies)
Brief Title: Scalar Closed Loop Intraoperative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dennis Turner, M.D. (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Dennis Turner, M.D., Professor of Neurosurgery, Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00085076; UH3NS103468 (NIH)
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intraoperative Recording During DBS Implant Surgery (Other): Participants will be recruited and enrolled from individuals who have Parkinson's disease (PD) and who already are scheduled to undergo the planned deep brain electrode placement for treatment of their movement disorder. Intraoperative recordings of participants' neural signals will be made through the implanted deep brain electrode(s).
  Interventions: Device: IPG; RC+S

INTERVENTIONS:
Device: IPG; RC+S — We will measure the effects of varying stimulation parameters on the neural activity in subjects with Parkinson's disease (PD).

SUMMARY:
The purpose of this study is to measure neural activity during deep brain stimulation (DBS). There are two types of neural activity that we will record from DBS electrodes during this study: DBS local evoked potentials (DLEPs) and spontaneous, local field potentials (LFPs). We will measure the effects of varying stimulation parameters on both the neural activity and changes in motor symptoms -- bradykinesia and tremor -- in subjects with Parkinson's disease (PD). Correlating neural activity characteristics with changes in symptoms will improve our understanding of the mechanisms of action of DBS. This intraoperative study will specifically compare our ability to record neural activity using circuitry developed at Duke for this purpose [Kent et al, 2015] to a new, implanted pulse generator (IPG; RC+S) developed by Medtronic. These intraoperative studies will specifically test a preliminary version of the RC+S (that is not designed for implantation), and will lead to a clinical trial assessing the efficacy of the implantable RC+S IPG in PD patients once this device is available and approved for this trial.

DETAILED DESCRIPTION:
The investigator will measure DBS local evoked potentials (DLEPs) and/or local field potentials (LFPs) together with motor symptoms (tremor and/or bradykinesia) in response to deep brain stimulation (DBS). The study will be conducted in the operating room at Duke University Medical Center. Additional operating room costs will be covered by institutional resources at Duke. The study will be performed on subjects who are undergoing implantation of the DBS system during an awake, stereotactic procedure for PD.

The subject group will only include patients undergoing a DBS implant procedure for PD. The surgical procedure will proceed as needed for treatment of Parkinson's disease (PD), including implantation of the DBS electrode (one into STN or dual electrodes into STN and GPi/GPe) into the targeted regions of the brain. For this research, subjects will receive temporary (~45 min) percutaneous extensions to the DBS electrode(s) and DBS lead cannula after implantation. These temporary extensions will connect to both our Duke stimulation and recording system or the Medtronic RC+S test recording system, alternating as needed, to allow recording and direct comparison of neural DLEP responses and/or LFPs using the two different stimulation/recording systems. Details of the stimulation and recording system are provided in the Study Interventions section. After the study is completed, the second DBS electrode (if placed) and the temporary percutaneous extensions will be removed. Then, the ordinary clinical conduct of the procedure will continue for treatment of the patient's movement disorder.

The investigator will measure tremor and/or bradykinesia in persons with PD during DBS. Subjects will be familiarized with and able to practice the evaluation tasks before preparation for surgery. Further, they will be asked to discontinue use of dopaminergic and/or anti-tremor medications overnight prior to the study (as is the clinical routine), to reduce variability of motor symptoms due to the time course of medications. The investigator will conduct evaluations using unilateral stimulation, with the limb contralateral to the side of stimulation used for measurement of motor symptoms. Subjects may also be asked to rate any side effects that they experience on a 0 - 10 scale.

Contacts on the subject's DBS electrode will be used for stimulation and recording. The four DBS contacts are designated as 0-1-2-3 in the ventral-dorsal direction. For monopolar stimulation, a single contact will be used for cathodic stimulation (1- or 2-) and a conductive pad will be placed on the subject's skin, outside of the sterile field, to serve as the return electrode. The recording contacts will be two other contacts on the DBS lead. For bipolar stimulation, DBS pulses will be applied between two electrode contacts, and the recording contacts will be the two remaining free contacts. The stimulus waveform will be a charge-balanced biphasic pulse, with charge restricted to values below the limit set by the manufacturer, 30 µC/cm2. Another conductive pad will be placed on the subject to serve as the recording reference. For subjects undergoing the DBS implantation surgery, the DBS lead cannula or a surgical retractor normally placed at the cranial incision site may also be used as the recording reference or return electrode.

In subjects with tremor-dominant PD, the investigator will record both the tremor and DLEP and/or LFP responses from the DBS electrode. Several trials will be conducted with different stimulation amplitudes, frequencies (≤185 Hz), temporal patterns, and contact configurations. The stimulation amplitude will be less than that identified to be uncomfortable to the subject or that generates side effects, as determined by a neurologist and/or neurosurgeon during the initial testing phase following implantation. The different stimulation parameters will be delivered in randomized order, and the subject will be blinded to the parameters. Measurements will be made during 2-minute trials, in which stimulation will be off for the first minute of the trial, and on for the remaining minute. At 30 s into both the off (baseline) and on phases of the trial, tremor will be measured for 20 s. The neural activity will also be measured from the electrode during both the off and on phases. The total amount of time necessary for data collection will be about 45 minutes.

Tremor will be measured using an accelerometer taped to the back of the subject's hand, and with the wrist extended such that the hand is parallel to the forearm. The elbow may either be supported or unsupported, depending on which induces greater tremor (determined prior to any trials in each subject). Tremor as measured by an accelerometer correlates well with clinical tremor rating scales [Elble et al, 2006].

In subjects with Parkinson's disease who do not have dominant tremor symptoms, the investigator will record both bradykinesia testing responses and DLEP and/or LFP potentials. Several trials will be conducted with different stimulation amplitudes, mean frequencies (≤185 Hz), temporal patterns, and contact configurations. The maximum amplitude delivered will be determined as described as above. The different stimulation parameters will be delivered in randomized order, and the subject will be blinded to the parameters. Measurements will be made in 10-minute trials, in which stimulation will be off for the first five minutes of the trial, and on for the remaining five minutes. At approximately 90, 210 and 250 s into both the off (baseline) and on phases of the trial, bradykinesia will be measured for 20 s. The neural activity will also be measured from the electrode during both the off and on phases of the trial. The total amount of time necessary for data collection will be about 45 minutes.

For bradykinesia measurements, the subject will be instructed to press alternately the right and left buttons of a computer mouse with the index and middle finger of their hand as rapidly and regularly as possible. Bradykinesia will be measured as the timing of alternating finger presses, a validated test of bradykinesia [Taylor-Tavares et al., 2005].

Before DBS surgery, the subject's baseline pathological motor symptoms may be assessed in the pre-operative setting, to familiarize the patient with the task ahead of the implant procedure. Tremor or bradykinesia will be measured using the previously-described accelerometer measurement or the mouse click task, respectively. This task will take about 5 minutes, and will be performed in the DBS-off condition. No sedation will be administered until after this has been completed.

Following DBS surgery, the subject's pre-operative MRI and post-operative high-resolution CT scans may be used to determine the location of DBS electrode contacts within the brain. Placement of the electrode during DBS implant surgery will not be altered by the research study.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease (PD) patients who are scheduled to already undergo the planned deep brain electrode placement for treatment of their movement disorder at Duke University Medical Center.
* Able to understand the study and consent form, and interested in proceeding with research during the invasive brain surgery to receive a DBS system for treatment of PD.

Exclusion Criteria:

* Inability to execute the motor tasks during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Turner, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Recording During DBS Implant Surgery
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Recording During DBS Implant Surgery
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recorded Evoked Neural Signals From Deep Brain Stimulation (DBS) Electrodes During DBS for Parkinson's Disease.
Description: Measured by the ability to record neural activity through DBS electrodes using circuitry developed at Duke for this purpose and/or a new implantable pulse generator (IPG; RC+S) developed by Medtronic. These intraoperative studies will specifically test a preliminary version of the RC+S that is not designed for implantation.
Time Frame: End of procedure, approximately 45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Recording During DBS Implant Surgery
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Number of Participants With Recorded DBS Local Evoked Potentials (DLEPs).
Description: Measured by the ability to record DLEPs (changes in local electric field in response to DBS stimulation) through DBS electrodes using circuitry developed at Duke for this purpose and/or a new implantable pulse generator (IPG; RC+S) developed by Medtronic. These intraoperative studies will specifically test a preliminary version of the RC+S that is not designed for implantation. The DLEP recordings will be serially averaged with stimulus-triggering to remove random noise while preserving the evoked response.
Time Frame: End of procedure, approximately 45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Recording During DBS Implant Surgery
Number analyzed (Participants) | 5
Participants | 5

3. Secondary Outcome: Number of Participants With Recorded Spontaneous, Local Field Potentials (LFPs).
Description: Measured by the ability to record LFPs (electrical activity in the local region of the DBS electrode) through DBS electrodes using circuitry developed at Duke for this purpose and/or a new implantable pulse generator (IPG; RC+S) developed by Medtronic. These intraoperative studies will specifically test a preliminary version of the RC+S that is not designed for implantation.
Time Frame: End of procedure, approximately 45 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Recording During DBS Implant Surgery
Number analyzed (Participants) | 5
Participants | 4

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intraoperative Recording During DBS Implant Surgery
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Recording During DBS Implant Surgery (N=5)
somnolence (Nervous system disorders) | 1
infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Recording During DBS Implant Surgery (N=5)
hyperhidrosis (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03270657/Prot_SAP_000.pdf